CLINICAL TRIAL: NCT05114408
Title: The Influence of Prehabilitation on the Surgical Patients Condition
Brief Title: Trimodal Prehabilitation in Patients Undergoing Elective Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Gdansk (Other)
Collaborators: University Clinical Centre, Gdansk (Other); EIT Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PREHAB1
Record Dates: First submitted 2021-07-14; First posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Cardiac Complication; Perioperative Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trimodal prehabilitation (Experimental): Patients qualified for elective surgery that meet criteria for prehabilitation
  Interventions: Other: 4 week trimodal prehabilitation course

INTERVENTIONS:
Other: 4 week trimodal prehabilitation course — trimodal prehabilitation in mixed: stationary and "at-home" structure

SUMMARY:
Patients scheduled for elective surgery will undergo 4 week course of trimodal prehabilitation

DETAILED DESCRIPTION:
Patients with high surgical risk will participate in 4 week prehabilitation that will consist of 4 stationary sessions - one per week - comprised of: physiotherapy session, psychological session and nutritional advice. During first session each patient will receive an activity monitor and dedicated mobile app that will record his daily performance.

ELIGIBILITY:
Inclusion Criteria:

* Age > 70 and/or American Society of American Society of Anesthesiologists Physical Status Classification System (ASA) 3-4
* Unfit patients

Exclusion Criteria:

* physical condition that makes the patient is not able to perform rehabilitation exercises
* cardiac and respiratory instability or high risk of its occurrence
* inability to use electronic devices used in the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-06-07 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
6 minute walk test | baseline and pre surgery
  change in aerobic capacity
Yale Physical Activity Survey (YPAS) | baseline and pre surgery
  change in physical activity
self-perceived health status scale (36-Item Short Form Survey - SF36) | baseline and pre surgery
  change in self-perceived health status (0 - min, 100 - max self perceived health score)
Global Leadership Initiative on Malnutrition (GLIM) scale | baseline and pre surgery
  change in nutritional status - malnutrition diagnosed if one phenotypical and one etiological criteria are fulfilled
  Severity based on phenotypic criteria:
  1. minimal value (moderate malnutrition)
  2. max value (severe malnutrition)
Hospital Anxiety and Depression (HAD) scale | baseline and pre surgery
  change in psychological status: depression and anxiety criteria 0 points min score - low level od depression and anxiety 21 max score
motivation questionaire (MQ) | baseline and pre surgery
  change in patient's motivation
  0-10 0 - low motiwation 10 max motivation
Perceives stress - Perceived Stress Questionaire (PSS) | baseline and pre surgery
  stress level - 0 - min value - no perceived stress 20 - maximal preceived stress

SECONDARY OUTCOMES:
Number of Participants requiring reintervention during initial hospitalization | 3 months after surgery
ICU length of stay | 3 months after surgery
Total hospital length of stay | 3 months after surgery
Number of Patients requiring Emergency room visits and hospital readmissions | at 30 days
Number of Patients with postoperative complications | 3 month after surgery
  number and severity

OTHER OUTCOMES:
Patient concentration questionaire (P3CQ) | after prehabilitation course
  Patient experience:
  0 - worst (medical staff not concentrated on patient) 19 - best experience (full concentration on patients needs)
Staff engagement questionaire (ACT) | after recruitment
  Staff engagement
cost analysis | 3 months after surgery
Continuity of Care Questionaire (NCQ) | after prehabilitation course
  form 0 - 5 pints 0 - lack of continuity of care 5 - maximal continuitu of care

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinical Center in Gdansk - Departament of Anesthesiolog and Intensive cCre, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: No